CLINICAL TRIAL: NCT04247958
Title: A Prospective Single-Center Evaluation of SureForm™ Staplers in Robotic-assisted Colorectal Procedures
Status: Completed | Type: Observational
Sponsor: Intuitive Surgical (Industry)
Responsible Party: Sponsor
Other Study IDs: ISI-dVCR-003
Record Dates: First submitted 2020-01-10; First posted 2020-01-30 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Benign Colon Tumor; Malignant Colorectal Tumor; Benign Colorectal Neoplasm
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Robotic-assisted colorectal resection: Subjects with either a suspected or confirmed benign or malignant disease of the colon and rectum who are scheduled to undergo a robotic-assisted resection of the colon or rectum.
  Interventions: Procedure: Colorectal resection

INTERVENTIONS:
Procedure: Colorectal resection — Robotic-assisted resection of the colon or rectum in subjects with benign or malignant colon or rectal disease, where SureForm™ Staplers are utilized for transection and/or creation of anastomosis.

SUMMARY:
The primary objective of this study is to evaluate the performance of SureForm™ Staplers (60 and 45) for transection and/or creation of anastomosis during robotic-assisted colorectal procedures.

DETAILED DESCRIPTION:
This is a prospective, single-center observational study to evaluate the performance of SureForm™ Staplers during robotic-assisted resections of either ascending or transverse or descending or sigmoid colon or rectum. Subjects with either a suspected or confirmed benign or malignant disease of the colon and rectum who are scheduled to undergo a robotic-assisted resection of the colon or rectum will be asked to provide informed consent for their participation in the study.

The study will be conducted at one institution with two surgeons performing the colorectal procedures. The surgeons will be using either the da Vinci Xi or X Surgical System which ever they use as per their standard of care for the colorectal procedure. Stapling will be performed with SureForm™ Staplers and any of the reloads as per the surgeon's standard of care for the transection and/or creation of anastomosis during robotic-assisted colorectal procedures.

ELIGIBILITY:
Inclusion Criteria:

* The subject must be 18 years of age or older at the time of consent
* Subject undergoing robotic-assisted colorectal procedure for benign or malignant colon or rectal disease, where SureForm™Staplers are utilized for transection and/or creation of anastomosis

Exclusion Criteria:

* Subject has had prior neoadjuvant (chemotherapy and/or radiation) therapy
* Subject with active bacterial or fungal infection
* Subject is contraindicated for general anesthesia or surgery
* Subject is undergoing an emergency procedure
* Subject has other major concomitant procedures (e.g. hepatectomies, incisional ventral hernia repair, nephrectomies, hysterectomy) planned along with colorectal procedure.
* Subject has metastatic disease and/or subject has life expectancy of less than 1 year
* Subject is under an immunomodulatory or immunosuppressive regimen (e.g. transplant patient, steroid requirement) within 30 days prior to the planned surgical procedure
* Subject has history of coagulation or hematologic disorder
* Pregnant or suspect pregnancy
* The subject is unable to comply with the follow-up visit schedule
* Subject has perforated, obstructing or locally invasive neoplasm (T4b)
* Subject with inflammatory bowel disease
* Subject is mentally handicapped or has a psychological disorder or severe systemic illness that would preclude compliance with study requirements or ability to provide informed consent
* Subject belonging to other vulnerable population, e.g, prisoner or ward of the state

Intra-Operative Exclusion Criteria:

* Subjects who require extensive dissection to release adhesions or with advanced cancer which may result in anastomotic leak and/or bleeding unrelated to the stapler.
* Inadequate visualization making an endoscopic approach not feasible
* Anatomy determined intra-operatively to be unsuitable for minimally invasive surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subject undergoing robotic-assisted colorectal procedure for suspected or confirmed benign or malignant colon or rectal disease.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2020-01-30 (Actual); Primary Completion 2021-07-21 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Number of SureForm™ Stapler fires and reload colors | During the procedure
  The primary endpoint of the study is to assess the number of fires and reload colors of SureForm™ Staplers utilized for the transection and/or creation of anastomosis during robotic-assisted colorectal procedures.

SECONDARY OUTCOMES:
Incidence of peri-operative and short term outcomes | 30 days post-operative
  The secondary endpoint of the study is to assess the incidence of peri-operative and short term outcomes following transection and/or creation of anastomosis using SureForm™ Staplers during robotic-assisted colorectal procedures.

CONTACTS AND LOCATIONS:
Locations (1):
- Oklahoma Surgical Hospital, Tulsa, Oklahoma, United States